CLINICAL TRIAL: NCT02321826
Title: Better Night - Better Day: a Randomized Controlled Trial of Listening to Music for Improving Insomnia
Brief Title: Music for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M&I2015
Record Dates: First submitted 2014-12-10; First posted 2014-12-22 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-04

CONDITIONS: Insomnia; Sleep Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — Music Therapy; Sound Recordings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Music (Experimental): Listening to music for 45 minutes at bedtime
  Interventions: Behavioral: Music
- Audiobook (Active Comparator): Listening to audiobook for 45 minutes at bedtime
  Interventions: Behavioral: Audiobook
- Control (No Intervention): No intervention control group

INTERVENTIONS:
Behavioral: Music — Participants choice among 4 genres of music matched on music characteristics
  Arms: Music
Behavioral: Audiobook — Participants choice among 4 types of audiobooks
  Arms: Audiobook

SUMMARY:
The aim of this study is to determine the effect of listening to music on sleep quality (subjective and objective), daytime dysfunction and neurophysiological arousal in patients with insomnia.

DETAILED DESCRIPTION:
Sleep problems are highly prevalent in modern society and poor sleep is associated with impaired physical and mental health with large costs for both individuals and society. Pharmacological treatment is recommended only for short-term use, and there is a need to study promising drug-free aids to improve sleep. Furthermore, the mechanisms of insomnia are not well understood. In the present project we will investigate if listening to music can improve sleep quality in persons suffering from insomnia. We will use a randomized controlled trial design including both subjective and objective measures of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia diagnosis

Exclusion Criteria:

* Use of hypnotic medications
* Alcohol or substance abuse
* Pregnant or breastfeeding women
* Sleep apnea with an apnea hypopnea index (AHI) >15
* Clinically significant restless leg syndrome or periodic limp movement disorder (PLMS>25)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-04; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Change in insomnia severity | Baseline and three-weeks follow-up
  Measured with the Insomnia Severity Index (ISI)
Change in subjective sleep quality | Baseline and three-weeks follow-up
  Measured with the Pittsburgh Sleep Quality Index (PSQI)

SECONDARY OUTCOMES:
Change in objective sleep quality (PSG) | Baseline and three-weeks follow-up
  Total sleep time, Sleep efficiency, sleep onset latency and wake after sleep onset as measured with polysomnography
Change in objective sleep quality (actigraphy) | Baseline and three-weeks follow-up
  Total sleep time, Sleep efficiency, sleep onset latency and wake after sleep onset as measured with actigraphy
Change in daytime dysfunction | Baseline and three-weeks follow-up
  Measured with the Fatigue severity scale (FSS), Becks Depression inventory (BDI-II), State-Trait Anxiety Inventory (STAI) and WHOQOL-BREF
Change in physiological arousal | Baseline and three-weeks follow-up
  Measured with ECG and respiration rate

CONTACTS AND LOCATIONS:
Overall Officials: Kira V Jespersen, Principal Investigator — Center of Functionally Integrative Neuroscience, Aarhus University
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No